CLINICAL TRIAL: NCT07089134
Title: Efficacy of Immersive Virtual Reality Rehabilitation on Patient Satisfaction and Experience, Functional and Clinical Outcomes, and Its Feasibility in Intensive Care Unit Treatment: a Randomized Controlled Trial
Brief Title: Virtual Reality in Intensive Care Unit: Patient Satisfaction, Clinical and Functional Outcomes, Feasibility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sirio-Libanes (Other)
Responsible Party: Principal Investigator, Wellington Yamaguti, Principal Investigator, Hospital Sirio-Libanes
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSL SP 2025-64
Record Dates: First submitted 2025-05-26; First posted 2025-07-28 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Hospitalized Patients; ICU Hospitalization; Intensive Care Unit-acquired Weakness
Keywords: virtual reality; rehabilitation; intensive care; stress; satisfaction; patient experience
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: Considering that patients enrolled in the study must complete a total of 6 to 14 rehabilitation protocol sessions, and in order to ensure the accuracy of the outcomes analyzed, participants who are absent for more than two consecutive rehabilitation sessions or who do not complete at least 70% of the total number of sessions will be excluded from the final analysis of the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traditional physiotherapy rehabilitation (Active Comparator): The traditional physiotherapeutic rehabilitation protocol will be guided by the characteristics of the early rehabilitation protocol in the ICU, structured by the rehabilitation service of Hospital Sírio-Libanês. This protocol provides recommendations for effective and applicable exercises based to the clinical reality, serving as a guiding resource in the care of critically ill patients.
  Interventions: Procedure: reabilitação fisioterapêutica tradicional
- physiotherapy using immersive virtual reality (Experimental): The immersive virtual reality physiotherapeutic rehabilitation protocol will employ 3D virtual reality headset that simulate human sensory input to create an immersive environment.
  Interventions: Procedure: fisioterapia utilizando realidade virtual imersiva

INTERVENTIONS:
Procedure: reabilitação fisioterapêutica tradicional — Active and passive exercises, and walking
  Arms: traditional physiotherapy rehabilitation
Procedure: fisioterapia utilizando realidade virtual imersiva — Use of immersive virtual reality headset for rehabilitation sessions
  Arms: physiotherapy using immersive virtual reality

SUMMARY:
Background: Virtual reality is recognized as a progressive technology with the potential to enhance the rehabilitation process. Immersive virtual reality-based treatments can improve motor outcomes in physical rehabilitation, reduce stress caused by the intensive care unit environment and maximize patients' recovery processes.

Objective: To analyze the efficacy of rehabilitation using immersive virtual reality on patient satisfaction and experience, functional and clinical outcomes and the feasibility of its application during the hospitalization period in an intensive care unit (ICU).

Methods: This is a randomized controlled clinical trial involving ICU patients aged 18 years or older, with an estimated ICU stay of ≥ 72 hours, the ability to understand and follow verbal instructions and no diagnosis of psychotic disorders, visual impairment, or hearing loss. Patients will be divided into two groups: one undergoing traditional physiotherapy rehabilitation - control group (CG), and the other receiving physiotherapy using immersive virtual reality (IVR group). The following evaluations will be conducted: mobility condition, physical and psychological discomfort, estimated physical activity level, occurrence of delirium, cognitive decline screening, functionality classification, motivation level, patient experience, sense of immersion in the virtual reality environment, patient satisfaction during the rehabilitation process, occurrence of adverse events, and protocol feasibility. Data will be presented in graphs and tables. Results will be considered statistically significant at a 5% significance level (p ≤ 0.05), and all analyses will be performed using SPSS Statistics version 22.

Expected results: The investigators expect to find evidence that rehabilitation using immersive virtual reality can promote and enable a more pleasant and less traumatic experience during the patient's hospitalization, with greater satisfaction and adherence to the proposed rehabilitation, in addition to being an effective tool to optimize patients' functional and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 years
* Glasgow Coma Scale (GCS) score ≥14
* Richmond Agitation-Sedation Scale (RASS) score between -1 and +1
* Negative for delirium according to the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU)
* Estimated ICU stay of ≥72 hours
* Able to communicate in Portuguese
* Understand and follow verbal instructions
* Have no psychotic disorders, visual impairment or hearing loss.

Exclusion Criteria:

* Hemodynamic instability
* Signs of respiratory distress
* Contact isolation for infectious diseases
* Conditions that limit head and neck movement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction | Day 1 and day 7 or intensive care unit discharge
  To assess patient satisfaction, the investigators will use the Net Promoter Score (NPS) method, it is a methodology that indicates the likelihood of a consumer recommending products or services to others. The results are interpreted using the following parameters: 75-100% is considered "excellent," 50-74% is classified as "very good" and below 49% as "poor."
Patient experience: Perceived workload | Day 1 and day 7 or intensive care unit discharge
  To evaluate patient experience, the Raw Task Load Index (RTLX) will be used to assess perceived workload during or immediately after rehabilitation sessions. It is a multidimensional scale scored from 0 to 100, with higher scores indicating greater cognitive load.
Patient experience: Perceived motivation | Day 1 and day 7 or intensive care unit discharge
  Perceived motivation will be assessed using the Intrinsic Motivation Inventory (IMI), a 7-point Likert scale evaluating the individual's subjective experience during an activity (1 = strongly disagree; 7 = strongly agree).
Patient experience: Perceived presence | Day 1 and day 7 or intensive care unit discharge
  Patients in the immersive virtual reality group will also complete the Presence Questionnaire (PQ), a self-report tool that measures perceived presence in the VR environment across four domains: Engagement, Immersion/Adaptation, Sensory Fidelity, and Interface Quality. The PQ uses a 5-point Likert scale, with higher scores reflecting a stronger sense of presence.

SECONDARY OUTCOMES:
Classification of physical activity level | Baseline
  Physical activity assessment will be conducted using the International Physical Activity Questionnaire (IPAQ). The short version consists of seven open-ended questions, allowing estimation of the time spent per week in different dimensions of physical activity (walking, moderate and vigorous activities) and physical inactivity (sitting time). Based on IPAQ scoring guidelines, patients can be classified as: very active, active, irregularly active, or sedentary.
Muscle Strength | Baseline and after 7 days or intensive care unit discharge
  Muscle strength will be assessed using the Medical Research Council (MRC) manual muscle test. This evaluation involves testing key upper limb muscles (shoulder abduction, elbow flexion, wrist extension) and lower limb muscles (hip flexion, knee extension, ankle dorsiflexion) against the examiner's resistance. Strength is rated on a scale from 0 (no muscle activation) to 5 (full range of motion against full examiner resistance). Classification is based on the degree of muscle contraction or range of motion for each muscle evaluated. The total score ranges from 0 (complete tetraparesis) to 60 points (normal muscle strength).
Mobility Assessment | Baseline and after 7 days or intensive care unit discharge
  Patient mobility will be assessed using the ICU Mobility Scale. This scale ranges from 0 to 10 within a single domain, where a score of 0 indicates very low mobility (e.g., the patient performs only passive exercises in bed), and a score of 10 indicates high mobility (e.g., the patient walks independently without assistance).
Functionality Classification | Baseline and after 7 days or intensive care unit discharge
  The International Classification of Functioning, Disability and Health (ICF) will be used to describe functionality and disability related to health conditions, considering body functions and structures, activity limitations, and participation restrictions in the patient's environment. A customized checklist adapted to the ICU context of Hospital Sírio-Libanês will be used in this study. Qualifiers specify the level of functioning, ranging from 0 (no impairment) to 4 (complete impairment). Codes 8 and 9 indicate lack of information or not applicable. In the body structure category, three qualifiers are used to describe the nature of the impairment. In the activity and participation category, two qualifiers are used: performance and capacity. For environmental factors, a positive score (1 to 4) indicates facilitators, while a negative score (-1 to -4) indicates barriers.
Delirium Assessment | Up to 7 days or intensive care unit discharge
  The diagnosis and monitoring of delirium during ICU stay will be performed using the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). This is a quick and accurate tool for diagnosing delirium in critically ill patients, combining sedation and delirium monitoring.
Cognitive Function Assessment | Baseline and after 7 days or intensive care unit discharge
  Cognitive functions will be assessed using the Montreal Cognitive Assessment (MoCA), a brief screening tool that evaluates a wide range of cognitive domains, including executive functions, visuospatial abilities, naming, memory recall, digits, sentence repetition, abstract reasoning, and orientation. MoCA is considered effective for detecting mild cognitive impairment and dementia. The test is simple and quick to administer, taking approximately 20 minutes. The maximum score is 30 points, with a cutoff of 26; scores above 26 are considered normal.
Assessment of Pain and Psychological Variables | Baseline and after 7 days or intensive care unit discharge
  To assess discomfort, the Numeric Rating Scale (NRS) will be used. This is a unidimensional tool that measures discomfort intensity and is suitable for conscious and communicative adult patients. Assessments will be performed before and after the rehabilitation protocol.
  For pain assessment, patients will be asked to rate their pain on a scale from 0 to 10, where 0 represents no pain and 10 indicates the worst possible pain.
  The same scale will be used to evaluate the perception of anxiety and stress, quantifying the intensity of these psychological variables.
Rehabilitation Protocol Feasibility | After 7 days or intensive care unit discharge
  The feasibility of the protocol will be measured through the adherence rate to immersive virtual reality therapy sessions. Adherence will be calculated as a percentage (%) using the formula: number of rehabilitation sessions completed / total number of eligible sessions × 100. In this study, a value above 70% will be considered indicative of good feasibility of the rehabilitation protocol.
Adverse Events: Fall risk | Up to 7 days or intensive care unit discharge
  Fall risk will be assessed using the Johns Hopkins Fall Risk Assessment Tool. This scale stratifies and establishes personalized preventive measures for hospitalized patients. The total score categorizes patients as low risk (0-5 points), moderate risk (6-13 points), or high risk (14-35 points).
Adverse Events: Presence of symptoms | Up to 7 days or intensive care unit discharge
  The presence of symptoms will be evaluated using the Simulator Sickness Questionnaire (SSQ), which assesses the presence and intensity of 16 symptoms, including general discomfort, fatigue, headache, eye strain, difficulty focusing, increased salivation, sweating, nausea, poor concentration, "heavy head," blurred vision, dizziness (eyes open/closed), vertigo, abdominal discomfort, and belching. Symptom intensity is rated as 0 (none), 1 (mild), 2 (moderate), or 3 (severe).

CONTACTS AND LOCATIONS:
Overall Officials: Wellington Yamaguti, PHD, Principal Investigator — Hospital Sírio-Libanês
Locations (1):
- Hospital Sírio Libanês, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No